CLINICAL TRIAL: NCT01018238
Title: A Multiple Dose, Randomised, Double-blind, Placebo-controlled, Multiple Site Study of Anti-C5a Receptor Antibody (NNC 0151-0000-0000) in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: An Investigation of NNC 0151-0000-0000 in Subjects With Systemic Lupus Erythematosus (SLE)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: See detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN8209-3608; U1111-1112-1881 (Other: WHO)
Record Dates: First submitted 2009-11-16; First posted 2009-11-23 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Inflammation; Systemic Lupus Erythematosus
MeSH Terms: conditions — Inflammation; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo arm (Placebo Comparator)
  Interventions: Drug: placebo
- Cohort 1 (Experimental)
  Interventions: Drug: NNC 0151-0000-0000
- Cohort 2 (Experimental)
  Interventions: Drug: NNC 0151-0000-0000
- Cohort 3 (Experimental)
  Interventions: Drug: NNC 0151-0000-0000
- Cohort 4 (Experimental)
  Interventions: Drug: NNC 0151-0000-0000

INTERVENTIONS:
Drug: NNC 0151-0000-0000 — Multiple doses in the range of 0.05mg/kg to 0.30mg/kg administered subcutaneously (under the skin)
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: placebo — Multiple doses of placebo (no active ingredients) administered subcutaneously (under the skin)
  Arms: Placebo arm

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this clinical trial is to investigate the safety, tolerability, pharmacokinetics and signs of bioactivity of increasing repeated doses of NNC 151-0000-0000 in subjects with Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
The trial was terminated before any patients were exposed to the trial drug based on new findings indicating that dose escalation with multiple doses should be performed in a different trial population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus (SLE)
* Disease duration: 6 months or longer
* Stable, mild to moderately active systemic lupus erythematosus (SLE)
* Receiving stable maintenance therapy

Exclusion Criteria:

* Significant Lupus Nephritis
* Active central nervous system (CNS) disease
* Significant arterial or venous thrombosis (blood clots) within 12 months prior to trial start
* Body weight of 260 lbs/120 kg or more
* History of alcohol or substance abuse
* History of cancer
* Infections
* Viral infections: HIV, Hepatitis B or C, Epstein-Barr Virus (EBV), Cytomegalovirus (CMV), Varicella-Zoster Virus (VZV), or Herpes Simplex Virus (HSV-1 or HSV-2)
* Tuberculosis
* Severe systemic bacterial, viral or fungal infections within the past 12 months prior to trial start
* Immunosuppressive and immune modulating therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Observed adverse events | From day -28 to day 113

SECONDARY OUTCOMES:
Number of adverse Events (including injection site reactions) | Every visit through study completion (Day 113)
Pharmacokinetics: terminal half-life, trough values, serum concentrations | Day 1 through Day 113
Pharmacodynamics: levels of serum, plasma, and urine markers, auto-antibodies | Day 1 through Day 113
Clinical disease endpoints: Systemic Lupus Erythematosus Disease Activity Index (SLEDAI), British Isles Lupus Assessment Group (BILAG), and Quality of Life by use of SF-36 (QOL) | Day 1 through Day 113

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Lake Success, New York, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com